CLINICAL TRIAL: NCT01058837
Title: Sudden Cardiac Death in Heart Failure Trial 10 Year Follow-up (SCD-HeFT 10 Year)
Brief Title: SCD-HeFT 10 Year Follow-up
Acronym: SCD-HeFT10 Yr
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Seattle Institute for Cardiac Research (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Abbott Medical Devices (Industry)
Responsible Party: Gust H. Bardy, MD; Principal Investigator, Seattle Institute for Cardiac Research
Other Study IDs: 1RC1HL100625 (NIH)
Record Dates: First submitted 2010-01-26; First posted 2010-01-29 (Estimated); Last update posted 2010-02-11 (Estimated); Status verified 2010-02

CONDITIONS: Left Ventricular Systolic Dysfunction; Congestive Heart Failure; Ischemic and Non-ischemic Cardiomyopathy; Sudden Cardiac Death Primary Prevention
Keywords: Sudden Cardiac Death; Implantable Cardioverter Defibrillator; Ventricular Fibrillation
MeSH Terms: conditions — Ventricular Dysfunction, Left; Heart Failure; Ischemia; Death, Sudden, Cardiac; Ventricular Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
No clinical trial that has examined the role of implantable cardioverter defibrillator (ICD) therapy in the prevention of Sudden Cardiac Death (SCD) has provided outcome data for longer than a few years. The NHLBI sponsored and placebo-controlled Sudden Cardiac Death in heart Failure Trial (SCD-HeFT) conducted from 1997 to 2003 had the largest number of patients and the longest average follow-up at 45.5 months. This study changed the national reimbursement policy for ICD therapy and remains the reference point for all other ICD evaluations in patients with congestive heart failure from ischemic or non-ischemic systolic dysfunction. Despite the outcome, the role of ICD therapy in the management of patients with heart failure has been questioned because of four principal concerns: numbers needed to treat to save a life, lead integrity over time, the negative consequences of shock therapy, and the cost of therapy. The purpose of this trial is to track down the remaining patients for a one-time follow-up regarding key outcome data.

DETAILED DESCRIPTION:
Long-term outcome data for implantable cardioverter defibrillator (ICD) therapy is sorely needed. We will acquire these data by re-approaching the patient population from the original Sudden Cardiac Death in Heart Failure Trial (SCD-HeFT).[Bardy 2005] This research is supported by the National Heart Lung and Blood Institute of the National Institutes of Health.

SCD-HeFT was originally conducted from 1997 to 2003. It demonstrated unequivocally that ICD's save lives in patients with heart failure compared to placebo or amiodarone. More than 26 peer-reviewed publications, including three NEJM papers, have resulted from this work.[Bardy 2005, Poole 2008, Mark 2008] Despite the quality of SCD-HeFT and the evidence of the life-saving ability of ICD therapy, the role of ICD therapy in the management of patients with heart failure continues to be questioned. This study will provide long-term follow-up of the SCD-HeFT patients, which will now exceed 10 years on average.

ELIGIBILITY:
Inclusion Criteria:

This is a one time follow-up on patients previously enrolled. -

Exclusion Criteria:

This is a one time follow-up on patients previously enrolled.

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: At the close of follow-up of the original SCD-HeFT study on October 31, 2003 there were a total of 666 deaths out of the enrollment population of 2521 patients. The American Recovery and Reinvestment Act (ARRA) of 2009 offers a perfect opportunity to do a one-time survey of the remaining 1855 patients from our last follow-up of October 31, 2003. Data on this population would allow us to obtain 10 year ICD follow-up data on the most detailed and largest ICD study ever done.
Sampling Method: Probability Sample
Enrollment: 1855 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-08 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
To compare 10-year mortality data on the remaining 1855 SCD-HeFT patients since the close of follow-up from October 31, 2003 in the 3 arms of the trial (ICD, placebo and amiodarone)based upon an intent-to-treat and an on-treatment analysis. | Two years

SECONDARY OUTCOMES:
To obtain outcome data in the major subgroups of SCD-HeFT: ischemic v. non-ischemic and NYHA Class II vs. Class III heart failure, and in woman and minorities. | Two years
To obtain 10-year ICD use rates (appropriate and inappropriate therapy), complication rates, lead failure rates and replacement rates. | Two Years
To validate or refute the observation that amiodarone increases mortality in NYHA Class III patients. | Two years
To obtain 10-year hospitalization and major procedure data. | Two years
To obtain 10-year quality of life data. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Gust H. Bardy, MD, Principal Investigator — Seattle Institute for Cardiac Research
Locations (1):
- Seattle Institute for Cardiac Research, Bellevue, Washington, United States

REFERENCES:
- [Background] Bardy GH, Lee KL, Mark DB, Poole JE, Packer DL, Boineau R, Domanski M, Troutman C, Anderson J, Johnson G, McNulty SE, Clapp-Channing N, Davidson-Ray LD, Fraulo ES, Fishbein DP, Luceri RM, Ip JH; Sudden Cardiac Death in Heart Failure Trial (SCD-HeFT) Investigators. Amiodarone or an implantable cardioverter-defibrillator for congestive heart failure. N Engl J Med. 2005 Jan 20;352(3):225-37. doi: 10.1056/NEJMoa043399. PMID 15659722
- [Derived] Poole JE, Olshansky B, Mark DB, Anderson J, Johnson G, Hellkamp AS, Davidson-Ray L, Fishbein DP, Boineau RE, Anstrom KJ, Reinhall PG, Packer DL, Lee KL, Bardy GH; SCD-HeFT Investigators. Long-Term Outcomes of Implantable Cardioverter-Defibrillator Therapy in the SCD-HeFT. J Am Coll Cardiol. 2020 Jul 28;76(4):405-415. doi: 10.1016/j.jacc.2020.05.061. PMID 32703511
- See also: Coordinating Center Website — http://www.sicr.org